CLINICAL TRIAL: NCT06224764
Title: Assessment of the Impact of the Return Home of Premature Newborns With Intrauterine Growth Retardation Weighing Less Than 2 Kilos (Low Birth Weight) on Short- and Long-term Morbidity/Mortality
Brief Title: Assessment of the Impact of the Return Home of Premature Newborns Less Than 2 Kilos Morbidity/Mortality
Acronym: Petit-Poids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRD1722; 2023-A02200-45 (Other: ANSM)
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Premature Birth
Keywords: Prematurity; Weight at discharge; Morbi-mortality; Neonatology
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Mother and Father questionnaires (on paper or by phone).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mother and Father questionnaires (Other): Mother and Father questionnaires (on paper or by phone) and data collectionon newborns weighing less than 2 kilos (at discharge from birth to 11 months)
  Interventions: Other: Mother and Father questionnaires

INTERVENTIONS:
Other: Mother and Father questionnaires — Mother and Father questionnaires (on paper or by phone) and data collectionon newborns weighing less than 2 kilos (at discharge from birth to 11 months)

SUMMARY:
The aim of this study is to evaluate the impact of discharge from hospital with a weight of less than 2 kilos.

To do this, the investigator will look at the short-term and long-term outcome of newborns weighing less than 2 kilos who were discharged from the neonatology department at the NOVO hospital between 2012 and 2024.

DETAILED DESCRIPTION:
Prematurity in itself, whether simple or associated with intrauterine growth retardation, continues to be a real public health problem. In addition to gestational age at birth, the presence of co-morbidities can affect the morbidity and mortality of premature babies, as well as the length of hospital stay.

Advances in neonatal care and the involvement and skills of parents in the care of premature infants have led to a considerable reduction in mortality among these patients. According to the latest recommendations published in November 2022 by the WHO, and thanks to changes in the criteria for discharging these patients in recent years, the same applies to low-birthweight infants.

The early and well-planned discharge of premature babies is currently the subject of a great deal of study and research. According to these studies, it has been shown that the essential criteria for this discharge are the physiological capacities and skills of these vulnerable patients (thermoregulation, autonomous feeding and breathing, etc.). Essential care, parental support and home visits by qualified health workers (PMI, HAD, etc.) are also essential.

Premature birth has a real impact on the economic consequences in several countries. Infants small for gestational age had longer hospital stays, were more likely to be admitted to an intensive care unit and were more likely to be hospitalised in the first year of life, resulting in higher costs.

It is against this backdrop that the NOVO hospital is proposing to evaluate the impact of discharging babies weighing less than 2 kilos. To do this, the investigator will base his study on the short-term and long-term outcome of newborns weighing less than 2 kilos who were discharged from the NOVO hospital's neonatology department between 2012 and 2024.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn baby (born at less than 37 days' gestation)
* Newborn baby with IUGR (Intra-Uterine Growth Retardation)
* Newborn baby hospitalised in the neonatology department of the NOVO hospital - Pontoise site
* Patient born between 01/01/2012 and 31/12/2024.
* Newborn who has left the neonatology department or the Kangaroo Unit to return home weighing less than 2 kg.
* Newborn beneficiary of a social security scheme or entitled person.

Exclusion Criteria:

* Newborn transferred to another hospital before discharge.
* Refusal by one of the parents.
* Parent does not speak or understand French.

Ages: 1 Month to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Observation of the short-term outcome of neonates discharged from the neonatology department hospital (Pontoise site) between 2012 and 2024 with a weight of less than 2 kilos. | At the end of the study, an average of 11 month
  The short-term outcom is observed with the number of newborns weighing less than 2 kilos readmitted to hospital 30 days after discharge from the neonatology department of the NOVO hospital (Pontoise site) between 01/01/2012 and 31/12/2024. This data will be obtained from the questionnaire sent to the child's parents (question number 9 - "At the time of discharge" section).

SECONDARY OUTCOMES:
Observation of weight growth | At the end of the study, an average of 11 month
  Z-score measurement for weight. Measured at systematic visits at 2 months, 4 months and 11 months.
Observation of height growth | At the end of the study, an average of 11 month
  Z-score measurement for height. Measured at systematic visits at 2 months, 4 months and 11 months.
Observation of the growth of the cranial perimeter | At the end of the study, an average of 11 month
  Z-score measurement for cranial perimeter. Measured at systematic visits at 2 months, 4 months and 11 months.
Observation of morbidity associated with neonatal discharge at less than 2 kilos | At the end of the study, an average of 6 month
  The morbidity is observed with the number of newborns with the following morbidities at 6 months post-discharge: digestive disorders (GERD, constipation, colic, blood in stools), feeding difficulties, bronchiolitis, infant asthma, hospital admissions and emergency room visits for all reasons, poor weight gain, secondary infection (questions number 10 and 11 in the questionnaire).
Observation of the incidence of Sudden Unexplained Infant Death Syndrome (SUIDS) | At the end of the study, an average of 11 month
  Number of Sudden Unexplained Infant Deaths Syndrome (SUIDs) at 11 months from discharge (question number 14) when the parent questionnaire is returned, supplemented by a call from the investigator to the parents if the patient has died, in order to find out whether he or she has suffered a Sudden Unexplained Infant Death Syndrome (SUIDS). This information will also be sought in the patient's medical records.
Remote observation of parents' experiences | At the end of the study, an average of 6 month
  Description of parental stress and worries about returning home, studied using a questionnaire created for the research and given to parents (stress before discharge: questions number 4, 7, 9 and 10 of the questionnaire, stress on returning home: questions number 7 and 13).
Observation of the support offered to parents | At the end of the study, an average of 6 month
  Description of the type of follow-up (HAH nurse, referring doctor, Day Hospital follow-up) organised on discharge This information will be obtained from the questionnaire asked of the parents of the patients concerned (question number 3 on return).
Description of medical positions on minimum discharge weight | At the end of the study, an average of 6 month
  Description of medical positions on minimum discharge weight, via a questionnaire sent to doctors in various neonatal intensive care units/paediatric intensive care units in the Paris region (questions number 12, 13, 14 and 15).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Suzanne BORRHOMEE, Principal Investigator — Hôpital NOVO
Locations (1):
- Resuscitation and neonatal medicine department - Hôpital NOVO - Pontoise site, Pontoise, France